CLINICAL TRIAL: NCT03088163
Title: The Value of DWI-MRI(Diffusion-weighted Imaging) in Evaluating the Early Efficacy of Liver Metastasis in Colorectal Cancer
Brief Title: The Value of Diffusion-weighted Imaging in Evaluating the Early Efficacy of Liver Metastasis in Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FDZL-MRinCLM
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: DWI-MRI
MeSH Terms: interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DWI-MRI (Experimental)
  Interventions: Device: Diffusion weighted magnetic resonance imaging

INTERVENTIONS:
Device: Diffusion weighted magnetic resonance imaging — The enrolled colorectal liver metastases patients will receive DWI-MRI screening to evaluate the liver metastases before the chemotherapy, after the first cycle of chemotherapy and in the regular efficacy evaluation time, respectively.
  Other Names: DWI-MRI

SUMMARY:
The study is designed to evaluate the value of DWI-MRI (Diffusion weighted magnetic resonance imaging) in predicting the efficacy of liver metastases after chemotherapy in colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years with histologically or cytologically confirmed advanced colorectal adenocarcinoma
* Eastern Cooperative Oncology Group performance status of 0 to 2
* life expectancy of ≥ 3 months
* at least one measurable liver metastatic lesion in MRI (≥10mm)
* have adequate bone marrow, hepatic, and renal function
* previously received no palliative chemotherapy

Exclusion Criteria:

* patients with previous chronic inflammatory bowel disease, chronic diarrhea or recurrent bowel obstruction
* patients with symptomatic brain metastases
* active clinical severe infection
* have contraindication of MRI screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2 months
  the response rate predicted by DWI-MRI

SECONDARY OUTCOMES:
Progression free survival | 2 months
Overall survival | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No